CLINICAL TRIAL: NCT00356200
Title: Ascending-Dose, Double-Blind, Placebo-Controlled, Bilateral Study of Intralesional Fluphenazine Decanoate in Psoriasis
Brief Title: Fluphenazine Decanoate for Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment criteria met
Sponsor: Tufts Medical Center (Other)
Collaborators: Immune Control (Industry)
Responsible Party: Alice B Gottlieb, MD, PhD, Tufts Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP-CL1
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — fluphenazine depot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluphenazine treated (Experimental): Treated with fluphenazine
  Interventions: Drug: Fluphenazine Decanoate
- Placebo (Placebo Comparator): Treated with Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluphenazine Decanoate — Fluphenazine decanoate marketed by APP Pharmaceuticals (25 mg/mL, 5 mL vial) was used in this study. This was an ascending dose study with the first cohort of 5 subjects dosed at 10 µg/mL, followed by 5 subject dosed in the second cohort at 100 µg/mL. Note: "APP Pharmaceuticals" is the name of the pharmaceutical company; APP is not an acronym.
  Arms: Fluphenazine treated
Drug: Placebo — The sterile placebo (sesame oil with 1.2% (w/v) benzyl alcohol) was prepared at the University of Iowa, Division of Pharmaceutical Services, a FDA registered pharmaceutical manufacturing facility.
  Arms: Placebo

SUMMARY:
We are doing this research study to evaluate the effectiveness and safety of fluphenazine decanoate when injected with a needle into psoriasis lesions in adults. Fluphenazine decanoate is FDA (U.S. Food and Drug Administration) approved for use in people who have schizophrenia and psychotic symptoms. Fluphenazine decanoate is not approved by the FDA for use in psoriasis. Fluphenazine decanoate slows T cell growth in cells in laboratory test tubes. Its usefulness and safety in people with psoriasis will be investigated in this study.

DETAILED DESCRIPTION:
Psoriasis is a hyperproliferative, inflammatory, immune-mediated skin disease that affects approximately 2% of the United States and European populations (Tutrone 2001, Kipnis 2005). This disease manifests as red, scaly plaques that are itchy and/or painful. Patients with psoriasis may be socially stigmatized because of their appearance. Currently, there is no cure for this condition. Often, repeated medical treatments are necessary and can become expensive. Treatment with topical corticosteroids is the mainstay therapy for mild to moderate psoriasis. In more severe cases, systemic therapies (e.g., cyclosporine) and phototherapy (e.g., ultraviolet B (UVB) irradiation) are used. These treatments, however, are associated with toxicities or inconvenience. There is anecdotal evidence to suggest that antipsychotic drugs have a beneficial effect on psoriasis (Gupta 2001, 2003).

Fluphenazine is a phenothiazine antipsychotic drug. In vitro, fluphenazine kills activated human T cells under conditions that do not affect resting T cells (Immune Control Inc. data not shown). To determine the size of a therapeutic window for human peripheral blood mononuclear cells (PBMC)s, Immune Control Inc. performed the following experiments. First, phytohemagglutinin- (PHA)-activated cells were exposed to 2, 10, or 20 µM fluphenazine for 0, 18, 24, 36, 48, or 72 hours. Second, resting cells were exposed to identical fluphenazine concentrations for identical time periods, after which the drug was washed out of the cells, and the cells activated with PHA. In all cases, deoxyribonucleic acid (DNA) synthesis was measured by exposing the cells to tritiated thymidine, and measuring the incorporated nucleotide by scintillation counting. The data show that exposure of activated cells to 10 µM fluphenazine for 72 hours, or 20 µM fluphenazine for 36 hours, caused the death of virtually all of the activated cells. The ability of the resting cells to initiate DNA synthesis after activation, by contrast, was largely unaffected by these fluphenazine exposures. Although we cannot precisely control intralesional fluphenazine concentrations, we expect that injections of up to 1 mg fluphenazine decanoate will yield local concentrations that exceed 10 µM without significant systemic fluphenazine concentrations.

We propose that fluphenazine will suppress proliferating T-lymphocytes in psoriatic plaques in vivo and thus result in healing of plaques. The objective of this study is to assess the safety and biologic activity of intralesional injection of fluphenazine decanoate in adult subjects with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years of age with psoriasis, in general good health
* Must have symmetric target lesions approximately 2-4 cm in diameter on each side of the body (e.g., thighs) with baseline target lesion score of 6 or higher (scale of 0-12) for each target
* Women of childbearing potential must agree to use two forms of contraception for the duration of the study

Exclusion Criteria:

* Infliximab (Remicade) or alefacept (Amevive) within the past 6 months (24 weeks)
* Etanercept (Enbrel), efalizumab (Raptiva), adalimumab (Humira), or other tumor necrosis factor- (TNF)-alpha inhibitor within the past 3 months (12 weeks)
* Other systemic psoriasis therapies (e.g., methotrexate, cyclosporine, acitretin) or PUVA (psoralen plus ultraviolet A) within the past 4 weeks
* Ultraviolet B (UVB) or topical therapy (other than over the counter (OTC) moisturizers and shampoos) within the past 2 weeks (including topical corticosteroids, vitamin A and D analogues)
* Receipt of an investigational agent within the past 4 weeks
* Systemic corticosteroid therapy
* Inability to understand consent or comply with protocol
* Pregnancy, lactation, or unwillingness to use adequate birth control during the study
* Impaired hepatic function
* Known Human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS), hepatitis B/C
* Blood dyscrasia
* Epilepsy
* Tardive dyskinesia
* Excessive alcohol consumption
* Current use of selective serotonin reuptake inhibitors (SSRI), tricyclic, or norephinephrine reuptake inhibitor antidepressants or use within 6 weeks of beginning the study
* Concurrent use of anti-seizure drugs, with the exception of gabapentin for treatment of neuropathy
* Use of phenothiazine antipsychotics or anticholinergics
* Known allergy to fluphenazine decanoate or other phenothiazines
* Known allergy to parabens/para-aminobenzoic acid (PABA), benzyl alcohol, sesame oil or sesame seeds
* Clinically significant mitral valve disease
* Clinically significant and uncontrolled cardiovascular disease
* QTc >450 msec, or evidence of a clinically significant dysrhythmia on electrocardiography (ECG)
* Operator of heavy machinery
* Pheochromocytoma
* History of breast cancer
* History of seizure disorder
* Occupational exposure to organophosphate insecticides
* Parkinson's disease and other related movement disorders
* Lab abnormalities including:
* Alanine aminotranferease (ALT)/aspartate aminotransferase (AST) ≥ 2X upper limit of reference range
* Creatinine ≥ 1.5X upper limit of reference range
* Bilirubin ≥ 2X upper limit of reference range
* Absolute total lymphocyte or polymorphonuclear leucocyte count ≤ 1000/uL or ≥ 3X upper limit of ref range
* Platelets ≤ 80,000/uL
* Hemoglobin ≤ 8.0 g/dL
* Glucose ≥ 200 mg/dL
* Fasting blood sugar ≥ 126 mg/dL
* Concurrent use of drugs listed in Appendix F

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice B Gottlieb, MD, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts-New England Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Tutrone WD, Kagen MH, Barbagallo J, Weinberg JM. Biologic therapy for psoriasis: a brief history, II. Cutis. 2001 Dec;68(6):367-72. PMID 11775769
- [Background] Kipnis CD, Myers WA, Opeola M, Gottlieb AB. Biologic treatments for psoriasis. J Am Acad Dermatol. 2005 Apr;52(4):671-82. doi: 10.1016/j.jaad.2004.12.032. No abstract available. PMID 15793519
- [Background] Gupta MA, Gupta AK. Psychiatric and psychological co-morbidity in patients with dermatologic disorders: epidemiology and management. Am J Clin Dermatol. 2003;4(12):833-42. doi: 10.2165/00128071-200304120-00003. PMID 14640776
- [Background] Gupta MA, Guptat AK. The use of antidepressant drugs in dermatology. J Eur Acad Dermatol Venereol. 2001 Nov;15(6):512-8. doi: 10.1046/j.1468-3083.2001.00278.x. PMID 11843209

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 10 ug/ml Fluphenazine Decanoate: Receiving fluphenazine decanoate (10 ug/ml) in a target lesion on one side of the body and placebo in a lesion on the other side of the body.
- Cohort 2: 100 ug/ml Fluphenazine Decanoate: Receiving fluphenazine decanoate (100 ug/ml) in a target lesion on one side of the body and placebo in a lesion on the other side of the body.
Period: Cohort 1: 10 ug/ml
Arm/Group | Cohort 1: 10 ug/ml Fluphenazine Decanoate | Cohort 2: 100 ug/ml Fluphenazine Decanoate
Started | 5 | 0
Completed | 4 | 0
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Period: Cohort 2: 100 ug/ml (New Patients)
Arm/Group | Cohort 1: 10 ug/ml Fluphenazine Decanoate | Cohort 2: 100 ug/ml Fluphenazine Decanoate
Started | 0 | 5
Completed | 0 | 3
Not Completed | 0 | 2
Not completed — Lack of Efficacy | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 10 ug/ml Fluphenazine Decanoate | Cohort 2: 100 ug/ml Fluphenazine Decanoate | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.6 (11.70) | 38.8 (6.69) | 39.1 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Secondary Outcome: Change in Target Lesion Pruritus Visual Analog Scale (VAS) at Week 4 Compared to Baseline.
Description: Target lesion pruritus as measured by the Visual Analog Scale (VAS) from 0 to 100 mm at week 4 compared to baseline (with 0 being no pruritis and 100 being maximum pruritis).
Time Frame: Baseline to week 4
Population: all 5 patients per cohort completed the visit at week 4
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Cohort 1, 10 ug/ml Fluphenazine Treated Lesion: lesion receiving 10 ug/ml Fluphenazine decanoate (Cohort 1)
- Cohort 1, Placebo Treated Lesion: lesion treated with placebo (Cohort 1)
- Cohort 2, 100 ug/ml Fluphenazine Treated Lesion: lesion receiving 100 ug/ml Fluphenazine decanoate (Cohort 2)
- Cohort 2, Placebo Treated Lesion: lesion treated with placebo (Cohort 2)
Arm/Group | Cohort 1, 10 ug/ml Fluphenazine Treated Lesion | Cohort 1, Placebo Treated Lesion | Cohort 2, 100 ug/ml Fluphenazine Treated Lesion | Cohort 2, Placebo Treated Lesion
Number analyzed (Participants) | 5 | 5 | 5 | 5
mm | -30 (35.07) | -27.2 (34.69) | -18 (34.87) | -32.6 (31.81)

2. Primary Outcome: Change in Target Lesion Score at Week 4 Compared to Baseline
Description: Change in score from 0-14 of target lesion disease activity based on scaling, erythema, and induration as determined by a physician assessor at week 4 compared to baseline (with 0 being no disease activity and 14 being maximum disease activity).
Time Frame: Baseline to week 4
Population: all 5 patients per cohort completed the visit at week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cohort 1, 10 ug/ml Fluphenazine Treated Lesion: Cohort 1 10 ug/ml Fluphenazine decanoate treated lesion
- Cohort 1, Placebo Treated Lesion: Cohort 1 lesion treated with placebo
- Cohort 2, 100 ug/ml Fluphenazine Treated Lesion: Cohort 2 100 ug/ml Fluphenazine decanoate treated lesion
- Cohort 2, Placebo Treated Lesion: Cohort 2 lesion treated with placebo
Arm/Group | Cohort 1, 10 ug/ml Fluphenazine Treated Lesion | Cohort 1, Placebo Treated Lesion | Cohort 2, 100 ug/ml Fluphenazine Treated Lesion | Cohort 2, Placebo Treated Lesion
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | -1 (2.45) | -0.8 (2.68) | -0.4 (2.19) | -1.5 (2.40)

ADVERSE EVENTS:
Arm/Group | Cohort 1: 10 ug/ml Fluphenazine Decanoate | Cohort 2: 100 ug/ml Fluphenazine Decanoate
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 10 ug/ml Fluphenazine Decanoate (N=5) | Cohort 2: 100 ug/ml Fluphenazine Decanoate (N=5)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cold/sinus symptoms (Infections and infestations) | 2 (2) | 1 (1)
contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
contact lens irritation (Eye disorders) | 0 (0) | 1 (1)
cough (Infections and infestations) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
injection site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — local reaction, occurred in both fluphenazine treated and placebo treated lesions
itchy lesions (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — local reaction. In both cohort 1 patients, occurred in both fluphenazine treated and placebo treated lesions. In the cohort 2 patient, occurred in only fluphenazine treated lesion.
lesion pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — local reaction, occurred in only fluphenazine treated lesion
migraine (Nervous system disorders) | 0 (0) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
psoriatic lesion spreading (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — local reaction, occurred in both fluphenazine treated and placebo treated lesions in addition to other non target lesions.
sunburn (1st degree) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — local reaction
tired (Nervous system disorders) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No